CLINICAL TRIAL: NCT03800342
Title: Recovery, Fatigability, and Proteomic Response to Aerobic Exercise Training in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Mason University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VCO2-Proteomics
Record Dates: First submitted 2018-12-18; First posted 2019-01-11 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Adult; Fatigue
Keywords: recovery; proteomics; cardiorespiratory fitness; exercise; aerobic exercise training
MeSH Terms: conditions — Fatigue; Motor Activity

STUDY DESIGN:
Intervention Model Description: One arm, a single group of healthy individuals, will perform cardiopulmonary exercise testing pre and post an aerobic exercise training program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Healthy (Experimental): Healthy individuals will participate in two separate days of cardiopulmonary exercise testing (CPET) (separated by a minimum of two, maximum of 7 days apart) prior to starting the aerobic exercise training program (AET). Individuals will then complete a 4-5 week (4x/week x 17 sessions) continuous, high-intensity AET. Each training session will consist of cycling for 3-5 minutes to warm-up, 45 minutes at 70% of heart rate reserve (HRR-determined from pre-training CPET), and 5-10 minutes to cool down. Following the AET, individuals will repeat the two separate days of CPET performed pre-training.
  Interventions: Other: Aerobic Exercise Training

INTERVENTIONS:
Other: Aerobic Exercise Training — see arm/group description

SUMMARY:
The purpose of this protocol is to investigate the role of expired non-metabolic carbon dioxide in the relationship between fatigability and recovery and the response to aerobic exercise training in healthy individuals. Both fatigability and recovery are profoundly influenced by mitochondrial energetics which can be inhibited by ionic by-product accumulation during exercise. Buffering mechanisms of these fatigue-inducing ions releases non-metabolic carbon dioxide (CO2) that can be measured as expired CO2 (VCO2) during cardiopulmonary exercise testing (CPET), however the role of non-metabolic VCO2 in the relationship between fatigability and recovery has yet to be investigated.

Furthermore, this study aims to identify the how the patterns of proteins in healthy individuals respond to aerobic exercise training (e.g. stationary cycling) over approximately one month. The underlying mechanisms of recovery after physical activity, including mechanisms or biological pathways that could be highlighted by analysis of proteins in urine, could add to scientific knowledge regarding physical activity tolerance and potential exercise interventions. This knowledge could eventually assist with designing precise and personalized exercise interventions to improve physical activity performance.

The investigators hypothesize that 1) non-metabolic CO2 will be at least moderately associated with the inverse relationship between fatigability and recovery; and 2) highly active adults, compared to sedentary individuals, will exhibit differential proteomic patterns in response to an initial acute bout and subsequent repeated bouts of aerobic exercise.

DETAILED DESCRIPTION:
Subjects will be recruited from the greater Washington D.C. metro area by word of mouth, university classes, healthcare provider referral, social media posting, and by posted fliers. Healthy males and females as determined by the Physical Activity Readiness Questionnaire Plus (PARQ+) will qualify to participate, regardless of their fitness level. The study design and participation will be explained to those who are potentially interested in participating in the study. Individuals interested in participating as subjects will complete the PARQ+ and those answering "no" to all of the PARQ+ questions will qualify for inclusion. Those answering "yes" to one or more of the questions will be asked follow-up questions to determine if they meet inclusion/exclusion criteria. Subjects will then be consented and enrolled for participation.

Visit 1: Subjects meeting all inclusion criteria and no exclusion criterion will be consented and enrolled in the study. Subjects will then complete the International Physical Activity Questionnaire (IPAQ) to describe their current levels of physical activity. Height and weight measurements of the subject will also be taken. Subjects will then complete a standard peak cardiopulmonary exercise test (pkCPET) to volitional exhaustion with near infrared spectroscopy (NIRS) assessment of muscle oxygenation and microvascular reactivity, bioimpedance cardiographic (ZCG) assessment of cardiac output and stroke volume, and electrocardiographic (EKG) measurement of heart rate (HR) at rest and during exercise. After a 10-minute passive recovery period, subjects will perform an endurance based CPET (enCPET) at intensity of 70% of the peak wattage reached during the pkCPET, again to volitional exhaustion followed by a final 10-minute passive recovery period to conclude day one of testing.

Visit 2: Subjects will complete a submaximal square-wave test (swCPET) for measurement of oxygen on-kinetics. After a 10-minute recovery period, subjects will complete the same enCPET they performed during Visit 1 testing. This testing will again be followed by a 10-minute recovery period. EKG measurements of HR will be taken during exercise and rest periods. Subjects will receive a urine collection cup to be used prior to visit 3. Subjects will be asked to collect approximately 75-90 mL of urine on the morning of Visit 3 to provide upon arrival. Subjects will be asked to log food intake using the form described below for 48 hours, starting 24 hours prior to Visit 3.

Visits 3-19: On days 3-19, subjects will complete a continuous high intensity aerobic exercise training (AET) protocol. Subjects will warm up for approximately 5-minutes, exercise within their predetermined HR range for 45 minutes, followed by a 5-10 min recovery period. HR will be monitored using a Polar chest strap worn by the subject and a paired watch and the heart rate reading on the cycle ergometer monitored by the investigators. The entire training session will take approximately 60 minutes. Following Visit 3, subjects will be provided with a 2nd urine sample cup and asked to collect a "first-morning" urine sample (75-90mL) at home on the day after visit 3. Subjects will be asked to provide subsequent first-morning midstream urine samples at home on the morning of and the morning after visits 7, 11, 15, and 19 (10 total urine samples). Subjects will be provided with a copy of their initial food log and asked to repeat their nutritional intake for the same timeframe as the initial sample for each subsequent sample (24 hours prior to pre-exercise sample until post-exercise sample).

Visit 20: Subjects will repeat the same procedures performed at Visit 1 including a pkCPET, 10-minute recovery, enCPET, 10-minute recovery, in that order. NIRS, ZCG, and EKG again will be collected throughout both the active and recovery portions of the testing.

Visit 21: Subjects will repeat the same procedures performed on day two of testing including a swCPET, 10-minute recovery, enCPET, 10-minute recovery, in the order. EKG data will again be collected during the active and recovery portions of the testing.

ELIGIBILITY:
Inclusion Criteria:

* age 18-60
* body mass index > 19 to <35 kg/m2
* able to pedal leg cycle ergometer
* able to comprehend and speak English

Exclusion Criteria:

* diabetes mellitus
* significant pulmonary dysfunction (eg. chronic obstructive lung disease; interstitial lung disease)
* hypertension
* anemia
* stroke
* cancer (other than melanoma)
* cardiac, pulmonary, thyroid, autoimmune, musculoskeletal, neurological, metabolic bone, mitochondrial, hepatic, renal, and/or psychiatric disease
* abnormal blood lipids
* active substance abuse or cognitive impairment
* chronic infection requiring antiviral or antibiotic treatment
* taking any medications that may limit exercise capacity or the ability to adapt to aerobic exercise training
* previously or currently on anticoagulant therapy or therapeutic hormone replacement/supplementation (excluding birth control)
* pregnant
* smoking

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2019-01-22 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Non-metabolic VCO2 | pre and post 5 week (4 training sessions per week, 17 total sessions) aerobic exercise training protocol
  Correlate measures of non-metabolic carbon dioxide (as measured by the contribution of total expired non-metabolic VCO2) with the correlative relationship between fatigability (as measured by total time during an endurance CPET and on-kinetics during a constant square-wave CPET) and recovery (as measured by VO2 and VCO2 following maximal and submaximal CPET). Compare changes in measures of non-metabolic carbon dioxide (as measured by the contribution of total expired non-metabolic VCO2) and changes in oxygen consumption (as measured by VO2) pre and post exercise training.

SECONDARY OUTCOMES:
Urinary proteome | This outcome will be assessed at 10 time points per participant: each morning of visits 3,4,7,8,11,12,15,16,19, and 20. Data will be collected during these 5 weeks and at post-testing occurring the week following the end of training.
  Proteome of urine samples as measured by mass spectrometry

CONTACTS AND LOCATIONS:
Overall Officials: Andrew A Guccione, PT, PhD, DPT, Principal Investigator — George Mason University
Locations (1):
- George Mason University, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Booth FW, Roberts CK, Laye MJ. Lack of exercise is a major cause of chronic diseases. Compr Physiol. 2012 Apr;2(2):1143-211. doi: 10.1002/cphy.c110025. PMID 23798298
- [Background] Lee IM, Shiroma EJ, Lobelo F, Puska P, Blair SN, Katzmarzyk PT; Lancet Physical Activity Series Working Group. Effect of physical inactivity on major non-communicable diseases worldwide: an analysis of burden of disease and life expectancy. Lancet. 2012 Jul 21;380(9838):219-29. doi: 10.1016/S0140-6736(12)61031-9. PMID 22818936
- [Background] Pedersen BK, Saltin B. Exercise as medicine - evidence for prescribing exercise as therapy in 26 different chronic diseases. Scand J Med Sci Sports. 2015 Dec;25 Suppl 3:1-72. doi: 10.1111/sms.12581. PMID 26606383
- [Background] Moholdt TT, Amundsen BH, Rustad LA, Wahba A, Lovo KT, Gullikstad LR, Bye A, Skogvoll E, Wisloff U, Slordahl SA. Aerobic interval training versus continuous moderate exercise after coronary artery bypass surgery: a randomized study of cardiovascular effects and quality of life. Am Heart J. 2009 Dec;158(6):1031-7. doi: 10.1016/j.ahj.2009.10.003. PMID 19958872
- [Background] Mora S, Cook N, Buring JE, Ridker PM, Lee IM. Physical activity and reduced risk of cardiovascular events: potential mediating mechanisms. Circulation. 2007 Nov 6;116(19):2110-8. doi: 10.1161/CIRCULATIONAHA.107.729939. Epub 2007 Oct 22. PMID 17967770
- [Background] Booth FW, Laye MJ. The future: genes, physical activity and health. Acta Physiol (Oxf). 2010 Aug;199(4):549-56. doi: 10.1111/j.1748-1716.2010.02117.x. Epub 2010 Mar 24. PMID 20345416
- [Background] Santos-Parker JR, Santos-Parker KS, McQueen MB, Martens CR, Seals DR. Habitual aerobic exercise and circulating proteomic patterns in healthy adults: relation to indicators of healthspan. J Appl Physiol (1985). 2018 Nov 1;125(5):1646-1659. doi: 10.1152/japplphysiol.00458.2018. Epub 2018 Sep 20. PMID 30236049
- [Background] Collins FS, Patrinos A, Jordan E, Chakravarti A, Gesteland R, Walters L. New goals for the U.S. Human Genome Project: 1998-2003. Science. 1998 Oct 23;282(5389):682-9. doi: 10.1126/science.282.5389.682. PMID 9784121
- [Background] Jameson JL, Longo DL. Precision medicine--personalized, problematic, and promising. N Engl J Med. 2015 Jun 4;372(23):2229-34. doi: 10.1056/NEJMsb1503104. Epub 2015 May 27. No abstract available. PMID 26014593
- [Background] Cornwall J, Elliott JM, Walton DM, Osmotherly PG. Clinical Genomics in Physical Therapy: Where to From Here? Phys Ther. 2018 Sep 1;98(9):733-736. doi: 10.1093/ptj/pzy069. No abstract available. PMID 29893975
- [Background] Buford TW, Roberts MD, Church TS. Toward exercise as personalized medicine. Sports Med. 2013 Mar;43(3):157-65. doi: 10.1007/s40279-013-0018-0. PMID 23382011
- [Background] Davidsen PK, Turan N, Egginton S, Falciani F. Multilevel functional genomics data integration as a tool for understanding physiology: a network biology perspective. J Appl Physiol (1985). 2016 Feb 1;120(3):297-309. doi: 10.1152/japplphysiol.01110.2014. Epub 2015 Nov 5. PMID 26542523
- [Background] Magni R, Espina BH, Liotta LA, Luchini A, Espina V. Hydrogel nanoparticle harvesting of plasma or urine for detecting low abundance proteins. J Vis Exp. 2014 Aug 7;(90):e51789. doi: 10.3791/51789. PMID 25145492
- [Background] Whitham M, Parker BL, Friedrichsen M, Hingst JR, Hjorth M, Hughes WE, Egan CL, Cron L, Watt KI, Kuchel RP, Jayasooriah N, Estevez E, Petzold T, Suter CM, Gregorevic P, Kiens B, Richter EA, James DE, Wojtaszewski JFP, Febbraio MA. Extracellular Vesicles Provide a Means for Tissue Crosstalk during Exercise. Cell Metab. 2018 Jan 9;27(1):237-251.e4. doi: 10.1016/j.cmet.2017.12.001. PMID 29320704
- [Background] Keller P, Vollaard NB, Gustafsson T, Gallagher IJ, Sundberg CJ, Rankinen T, Britton SL, Bouchard C, Koch LG, Timmons JA. A transcriptional map of the impact of endurance exercise training on skeletal muscle phenotype. J Appl Physiol (1985). 2011 Jan;110(1):46-59. doi: 10.1152/japplphysiol.00634.2010. Epub 2010 Oct 7. PMID 20930125
- [Background] Hecksteden A, Kraushaar J, Scharhag-Rosenberger F, Theisen D, Senn S, Meyer T. Individual response to exercise training - a statistical perspective. J Appl Physiol (1985). 2015 Jun 15;118(12):1450-9. doi: 10.1152/japplphysiol.00714.2014. Epub 2015 Feb 5. PMID 25663672
- [Background] Lane RK, Hilsabeck T, Rea SL. The role of mitochondrial dysfunction in age-related diseases. Biochim Biophys Acta. 2015 Nov;1847(11):1387-400. doi: 10.1016/j.bbabio.2015.05.021. Epub 2015 Jun 4. PMID 26050974
- [Background] Lombardi A, Silvestri E, Cioffi F, Senese R, Lanni A, Goglia F, de Lange P, Moreno M. Defining the transcriptomic and proteomic profiles of rat ageing skeletal muscle by the use of a cDNA array, 2D- and Blue native-PAGE approach. J Proteomics. 2009 May 2;72(4):708-21. doi: 10.1016/j.jprot.2009.02.007. Epub 2009 Mar 5. PMID 19268720
- [Background] Wisloff U, Stoylen A, Loennechen JP, Bruvold M, Rognmo O, Haram PM, Tjonna AE, Helgerud J, Slordahl SA, Lee SJ, Videm V, Bye A, Smith GL, Najjar SM, Ellingsen O, Skjaerpe T. Superior cardiovascular effect of aerobic interval training versus moderate continuous training in heart failure patients: a randomized study. Circulation. 2007 Jun 19;115(24):3086-94. doi: 10.1161/CIRCULATIONAHA.106.675041. Epub 2007 Jun 4. PMID 17548726
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Oberg AL, Vitek O. Statistical design of quantitative mass spectrometry-based proteomic experiments. J Proteome Res. 2009 May;8(5):2144-56. doi: 10.1021/pr8010099. PMID 19222236
- [Background] Gemperline DC, Scalf M, Smith LM, Vierstra RD. Morpheus Spectral Counter: A computational tool for label-free quantitative mass spectrometry using the Morpheus search engine. Proteomics. 2016 Mar;16(6):920-4. doi: 10.1002/pmic.201500420. PMID 26791624
- [Background] Lavallee-Adam M, Rauniyar N, McClatchy DB, Yates JR 3rd. PSEA-Quant: a protein set enrichment analysis on label-free and label-based protein quantification data. J Proteome Res. 2014 Dec 5;13(12):5496-509. doi: 10.1021/pr500473n. Epub 2014 Oct 16. PMID 25177766
- [Background] Pascovici D, Handler DC, Wu JX, Haynes PA. Multiple testing corrections in quantitative proteomics: A useful but blunt tool. Proteomics. 2016 Sep;16(18):2448-53. doi: 10.1002/pmic.201600044. PMID 27461997
- [Background] Finsterer J, Mahjoub SZ. Fatigue in healthy and diseased individuals. Am J Hosp Palliat Care. 2014 Aug;31(5):562-75. doi: 10.1177/1049909113494748. Epub 2013 Jul 26. PMID 23892338
- [Background] Aaronson LS, Teel CS, Cassmeyer V, Neuberger GB, Pallikkathayil L, Pierce J, Press AN, Williams PD, Wingate A. Defining and measuring fatigue. Image J Nurs Sch. 1999;31(1):45-50. doi: 10.1111/j.1547-5069.1999.tb00420.x. PMID 10081212
- [Background] Eldadah BA. Fatigue and fatigability in older adults. PM R. 2010 May;2(5):406-13. doi: 10.1016/j.pmrj.2010.03.022. PMID 20656622
- [Background] Kim I, Hacker E, Ferrans CE, Horswill C, Park C, Kapella M. Evaluation of fatigability measurement: Integrative review. Geriatr Nurs. 2018 Jan-Feb;39(1):39-47. doi: 10.1016/j.gerinurse.2017.05.014. Epub 2017 Jun 27. PMID 28666548
- [Background] Keyser RE, Woolstenhulme JG, Chin LM, Nathan SD, Weir NA, Connors G, Drinkard B, Lamberti J, Chan L. Cardiorespiratory function before and after aerobic exercise training in patients with interstitial lung disease. J Cardiopulm Rehabil Prev. 2015 Jan-Feb;35(1):47-55. doi: 10.1097/HCR.0000000000000083. PMID 25313451
- [Background] Barbosa JF, Bruno SS, Cruz NS, de Oliveira JS, Ruaro JA, Guerra RO. Perceived fatigability and metabolic and energetic responses to 6-minute walk test in older women. Physiotherapy. 2016 Sep;102(3):294-9. doi: 10.1016/j.physio.2015.08.008. Epub 2015 Sep 28. PMID 26565376
- [Background] Keyser RE. Peripheral fatigue: high-energy phosphates and hydrogen ions. PM R. 2010 May;2(5):347-58. doi: 10.1016/j.pmrj.2010.04.009. PMID 20656616
- [Background] Nanas S, Nanas J, Kassiotis C, Nikolaou C, Tsagalou E, Sakellariou D, Terovitis I, Papazachou O, Drakos S, Papamichalopoulos A, Roussos C. Early recovery of oxygen kinetics after submaximal exercise test predicts functional capacity in patients with chronic heart failure. Eur J Heart Fail. 2001 Dec;3(6):685-92. doi: 10.1016/s1388-9842(01)00187-8. PMID 11738220
- [Background] Short KR, Sedlock DA. Excess postexercise oxygen consumption and recovery rate in trained and untrained subjects. J Appl Physiol (1985). 1997 Jul;83(1):153-9. doi: 10.1152/jappl.1997.83.1.153. PMID 9216958
- [Background] Belardinelli R, Lacalaprice F, Carle F, Minnucci A, Cianci G, Perna G, D'Eusanio G. Exercise-induced myocardial ischaemia detected by cardiopulmonary exercise testing. Eur Heart J. 2003 Jul;24(14):1304-13. doi: 10.1016/s0195-668x(03)00210-0. PMID 12871687
- [Background] Scrutinio D, Passantino A, Lagioia R, Napoli F, Ricci A, Rizzon P. Percent achieved of predicted peak exercise oxygen uptake and kinetics of recovery of oxygen uptake after exercise for risk stratification in chronic heart failure. Int J Cardiol. 1998 Apr 1;64(2):117-24. doi: 10.1016/s0167-5273(98)00019-9. PMID 9688429
- [Background] Thompson RB, Pagano JJ, Mathewson KW, Paterson I, Dyck JR, Kitzman DW, Haykowsky MJ. Differential Responses of Post-Exercise Recovery of Leg Blood Flow and Oxygen Uptake Kinetics in HFpEF versus HFrEF. PLoS One. 2016 Oct 4;11(10):e0163513. doi: 10.1371/journal.pone.0163513. eCollection 2016. PMID 27701422
- [Background] Fiedler GB, Schmid AI, Goluch S, Schewzow K, Laistler E, Niess F, Unger E, Wolzt M, Mirzahosseini A, Kemp GJ, Moser E, Meyerspeer M. Skeletal muscle ATP synthesis and cellular H(+) handling measured by localized (31)P-MRS during exercise and recovery. Sci Rep. 2016 Aug 26;6:32037. doi: 10.1038/srep32037. PMID 27562396
- [Background] Bower JE. Fatigue, brain, behavior, and immunity: summary of the 2012 Named Series on fatigue. Brain Behav Immun. 2012 Nov;26(8):1220-3. doi: 10.1016/j.bbi.2012.08.009. Epub 2012 Aug 31. PMID 22964543
- [Background] Vestergaard S, Nayfield SG, Patel KV, Eldadah B, Cesari M, Ferrucci L, Ceresini G, Guralnik JM. Fatigue in a representative population of older persons and its association with functional impairment, functional limitation, and disability. J Gerontol A Biol Sci Med Sci. 2009 Jan;64(1):76-82. doi: 10.1093/gerona/gln017. Epub 2009 Jan 27. PMID 19176328
- [Background] Schnelle JF, Buchowski MS, Ikizler TA, Durkin DW, Beuscher L, Simmons SF. Evaluation of two fatigability severity measures in elderly adults. J Am Geriatr Soc. 2012 Aug;60(8):1527-33. doi: 10.1111/j.1532-5415.2012.04062.x. Epub 2012 Aug 2. PMID 22860899
- [Background] Alexander NB, Taffet GE, Horne FM, Eldadah BA, Ferrucci L, Nayfield S, Studenski S. Bedside-to-Bench conference: research agenda for idiopathic fatigue and aging. J Am Geriatr Soc. 2010 May;58(5):967-75. doi: 10.1111/j.1532-5415.2010.02811.x. PMID 20722821
- [Background] Distefano G, Standley RA, Zhang X, Carnero EA, Yi F, Cornnell HH, Coen PM. Physical activity unveils the relationship between mitochondrial energetics, muscle quality, and physical function in older adults. J Cachexia Sarcopenia Muscle. 2018 Apr;9(2):279-294. doi: 10.1002/jcsm.12272. Epub 2018 Jan 24. PMID 29368427
- [Background] de Groote P, Millaire A, Decoulx E, Nugue O, Guimier P, Ducloux. Kinetics of oxygen consumption during and after exercise in patients with dilated cardiomyopathy. New markers of exercise intolerance with clinical implications. J Am Coll Cardiol. 1996 Jul;28(1):168-75. doi: 10.1016/0735-1097(96)00126-x. PMID 8752810
- [Background] Garcia-Saldivia M, Ilarraza-Lomeli H, Myers J, Lara J, Bueno L. Effect of physical training on the recovery of acute exercise, among patients with cardiovascular disease. Arch Cardiol Mex. 2017 Jul-Sep;87(3):199-204. doi: 10.1016/j.acmx.2016.11.004. Epub 2016 Dec 13. PMID 27979503
- [Background] Beaver WL, Wasserman K, Whipp BJ. A new method for detecting anaerobic threshold by gas exchange. J Appl Physiol (1985). 1986 Jun;60(6):2020-7. doi: 10.1152/jappl.1986.60.6.2020. PMID 3087938
- [Background] Brooks, G. A., Fahey, T. D. & Baldwin, K. M. Exercise physiology: human bioenergetics and its applications. (McGraw-Hill, 2005).